CLINICAL TRIAL: NCT03390283
Title: A Survey of Parent/Caregiver Practices on the Storage, Use, and Disposal of Opioids
Brief Title: A Survey of Parent/Caregiver Practices on the Storage, Use, and Disposal of Opioids in a Comprehensive Cancer Center
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2017-0396; NCI-2018-00986 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0396 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-12-28; First posted 2018-01-04 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Caregiver; Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (Online survey): Participants complete online survey on an iPad over 20 minutes.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Complete online survey

SUMMARY:
This trial uses a survey to study parent and caregiver practices on the storage, use, and disposal of opioids in a comprehensive cancer center. It is not known if parents and/or caregivers are aware of the guidelines and recommendations for proper and safe disposal of opioids. This survey will help health care providers assess the needs and improve the safety of patients and their families from the potential dangers of misuse and abuse of prescription opioid medications.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the frequency of unsafe storage, use, and disposal of unused and currently used opioids by parents and/or caregivers of patients 18 years and younger at MD Anderson Cancer Center.

II. To explore potential association between other covariates with the unsafe storage, use, and disposal of opioids.

OUTLINE:

Participants complete online survey on an iPad over 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* PARENTS/CAREGIVERS: Must be at least 18 years old (a. The child of the parents/caregivers must be 18 years old or younger; b. The child of the parents/caregivers must have received an opioid prescription within the last six months.)
* PARENTS/CAREGIVERS: Must be able to understand, read, write, and speak English.
* PARENTS/CAREGIVERS: Parent/caregiver must sign an informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Parents/caregivers of a child (under 18) who has received an opioid prescription within the last 6 months
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Reported frequencies of unsafe storage of opioids | Up to 2 years
  The unsafe storage of opioids is defined as having opioids in the open where anyone can see it, in a medicine cabinet that is not locked, or hidden but not locked. Will estimate the proportion along with a 95% confidence interval. The distribution of the primary outcome by demographic information will be presented in cross tabulations. The association between the primary outcomes and demographic information/other behavior will be explored by Chi-Squared test or Fisher's exact test when appropriate. Logistic regression models may be employed to assess the effect of demographic factors on the unsafe storage of opioids. Other statistics methods may be used when appropriate.
Reported frequencies of unsafe use of opioids | Up to 2 years
  This is defined as giving more opioid than prescribed to the child very frequently, frequently, occasionally, infrequently, or very infrequently. Will estimate the proportion along with a 95% confidence interval. The distribution of the primary outcome by demographic information will be presented in cross tabulations. The association between the primary outcomes and demographic information/other behavior will be explored by Chi-Squared test or Fisher's exact test when appropriate. Logistic regression models may be employed to assess the effect of demographic factors on the unsafe storage of opioids. Other statistics methods may be used when appropriate.
Reported frequencies of unsafe disposal of opioids | Up to 2 years
  This is defined as throwing unused pills in the trash without any modification. Will estimate the proportion along with a 95% confidence interval. The distribution of the primary outcome by demographic information will be presented in cross tabulations. The association between the primary outcomes and demographic information/other behavior will be explored by Chi-Squared test or Fisher's exact test when appropriate. Logistic regression models may be employed to assess the effect of demographic factors on the unsafe storage of opioids. Other statistics methods may be used when appropriate.

SECONDARY OUTCOMES:
Other covariates | Up to 2 years
  The association between unsafe storage, use and disposal and other variables including the presence of other children living in the home [defined as answering Question 9 as having minor children (age < 18 years) in the home], a family history of misuse of prescription drugs, street drugs or alcohol, a family history of psychiatric illness or other unsafe uses of opioid medications that do not relate directly to the child, such as if a caregiver takes or sells the child's medication will be analyzed. Demographic variables collected in the first part of the survey will be used to explore possible associations with unsafe storage, use or disposal of opioids.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Madden, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org